CLINICAL TRIAL: NCT06689917
Title: An Early Exploratory Clinical Study of the Safety, Tolerability and Preliminary Efficacy of JY231 Injection in the Treatment of Relapsed or Refractory B-cell Lymphoma/Leukaemia
Brief Title: JY231(JY231) Injection for the Treatment of Relapsed or Refractory B Cell Lymphoma/ Leukemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Jia Wei, professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JY-CT-24-001
Record Dates: First submitted 2024-11-10; First posted 2024-11-15 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: B-ALL; B-NHL

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JY231 injection for the treatment of relapsed or refractory B cell lympho Early exploratory clinica (Experimental): JY231 Injection for the Treatment of relapsed or refractory B cell lymphoma/ leukemia subjects who meet the inclusion criteria will receive intravenous JY231. JY231 infusion will produce CAR-T cells in the body.
  Interventions: Drug: JY231 Injection

INTERVENTIONS:
Drug: JY231 Injection — This study employs two pretreatment regimens:
  In the lymphodepletion regimen, upon enrollment, subjects undergo leukapheresis followed by 3-5 days of lymphodepleting therapy with fludarabine and cyclophosphamide, culminating in intravenous infusion of JY231 and autologous patient PBMCs via a double-lumen catheter; in the non-lymphodepletion regimen, subjects receive direct intravenous injection of the JY231 preparation immediately after enrollment.

SUMMARY:
This study is an investigator-initiated single center, single arm clinical study with a target population of patients with relapsed or refractory B cell lymphoma / leukemia. It is an early exploratory clinical study of the safety, tolerability and initial efficacy of JY231 injection in the treatment of relapsed or refractory B cell lymphoma / leukemia.

DETAILED DESCRIPTION:
This open-label, single-arm study is designed to evaluate the efficacy and safety of in vivo CAR-T cell therapy in patients with relapsed/refractory B-cell lymphoma/leukaemia. This study incorporates two pretreatment regimens: lymphodepletion and non-lymphodepletion.

In the lymphodepletion regimen:

Upon enrolment, leukapheresis will be performed. Subjects will then undergo 3-5 days of lymphodepleting therapy with fludarabine and cyclophosphamide, followed by concomitant intravenous infusion of the JY231 preparation and autologous peripheral blood mononuclear cell(PBMC) via a double-lumen catheter.

In the non-lymphodepletion regimen:

Patients will receive direct intravenous injection of the JY231 preparation.

Following infusion, subjects will undergo safety and efficacy assessments for up to 3 months. For those achieving sustained remission at 3 months post-infusion, follow-up will be conducted for at least 24 months to evaluate disease control status.

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily sign informed consent and are willing and able to comply with all trial requirements;
2. Age is 18-75 years old and gender is not limited;
3. Malignancy cells in bone marrow or peripheral blood are Cluster of Differentiation 19 - positive(CD19+) detected by flow cytometric analysis;
4. Meet the clinical criteria for relapsed or refractory B-cell lymphoma, including: indolent lymphoma (iNHL), such as follicular lymphoma (FL) and marginal zone lymphoma (MZL); aggressive B-cell lymphoma, like diffuse large B-cell lymphoma (DLBCL), primary mediastinal large B-cell lymphoma (PMBCL), transformed follicular lymphoma (TFL), and T-rich lymphocyte-bearing large B-cell lymphoma (TCRBCL), or have a diagnosis of acute B-lymphocytic leukemia (B-ALL) and meet one of the following conditions:

   * Refractory B-ALL: those who did not achieve complete remission after 2 courses of standard induction regimen chemotherapy, or those who did not achieve complete remission after first-line or multi-line salvage chemotherapy;
   * Relapsed B-ALL: relapse within 12 months after first remission, or relapse after first-line / multi-line salvage chemotherapy;
   * Relapse after autologous or allogeneic hematopoietic stem cell transplantation; In addition, patients with Philadelphia chromosome positive (Ph +) should be relapsed after at least two tyrosine kinase inhibitors (TKI) treatment, or they could not tolerate TKI therapy, or have a t315i mutation, resistant to TKI drugs.
5. Morphological examination of bone marrow cells showed the proportion of primitive and naive lymphocytes was> 5%;
6. No Hematopoietic Stem Cell Transplantation(HSCT) within 6 months before enrollment;
7. At least one measurable lesion was imaging for relapsed or refractory B cell lymphoma, long diameter of> 15mm, or extranodal lesion of> 10mm, along with a positive Positron Emission Tomography - Computed Tomography(PET-CT) examination.
8. More than 12 weeks of expected survival period
9. Baseline Eastern Cooperative Oncology Group(ECOG) score was 0-1;
10. Adequate organ function (criteria regarding liver and kidney function can be moderately relaxed):

    * Glutamic aminotransferase (ALT) ≤3 times upper limit of normal (ULN);
    * Grass aminotransferase (AST) ≤3 times ULN;
    * Total bilirubin ≤1.5 times ULN;
    * Serum creatinine ≤ 1.5 times ULN, or creatinine clearance ≥ 60 mL/min;
    * Indoor oxygen saturation ≥ 92%;
    * Left ventricular ejection fraction (LVEF)≥55%, echocardiography confirmed no pericardial effusion and no clinically significant ECG findings;
    * There is no clinically significant pleural effusion;
11. Adequate bone marrow reserve without transfusion, defined as:

    * Absolute neutrophil count (ANC)>1.000 / mm3;
    * Absolute lymphocyte count (ALC)≥ 300 / mm3;
    * Platelet≥50.000/mm3;
    * Hemoglobin>8.0 g/dl;
12. Subjects using the following drugs need to meet the following conditions:

    * Steroids: The therapeutic dose of steroids must be stopped 72 hours before JY231 infusion. However, physiological alternative doses of steroids are allowed;
    * Immunosuppression: Any immunosuppressive drug must be stopped at ≥4 weeks prior to enrollment;
    * Antiproliferative therapy other than lymphodepletion chemotherapy within two weeks of infusion;
    * Cluster of Differentiation 20(CD20) antibody-related therapy must be stopped within 4 weeks before infusion or 5 half-lives after the CD20 antibody;
    * CNS disease prophylaxis must be stopped 1 week before JY231 infusion (e. g. intrathecal methotrexate).
13. Reproductive men, sexual partners ensure effective contraception; fertile women, adopted effective contraception and agreed to use contraception throughout the study period.

Exclusion Criteria:

1. Subjects with active cerebrospinal fluid malignant cells or brain metastases, or subjects with active central nervous system (CNS) lymphoma, or CNS leukaemia;
2. Subjects with a history of active CNS disease, such as seizures, cerebrovascular ischemia / hemorrhage, dementia, cerebellar disease, or any autoimmune disease associated with CNS involvement;
3. Subjects who have received other study drugs within 30 days before screening, or are still in the washout period;
4. Patients who have previously received any anti-CD19 / anti-Cluster of Differentiation 3(CD3) therapy or any other anti-CD19 therapy (except for those with normal T cell numbers and function and with CD19-positive tumors);
5. Patients who have been previously treated with any gene therapy product, including Chimeric Antigen Receptor T(CAR-T) therapy (except patients who do not have CAR-T cells in vivo and have normal T cell number and function and are with CD19 positive tumors);
6. Subjects with radiation therapy within 2 weeks prior to the infusion;
7. Subjects with active hepatitis B (defined as Hepatitis B Virus(HBV) DNA test value> 500 IU / mL) or hepatitis C (HCV RNA positive); subjects with HIV positive or treponema pallidum positive;
8. Subjects with uncontrolled acute life-threatening bacterial, viral, or fungal infection (e. g. positive blood culture 72 hours before infusion);
9. Subjects with unstable angina pectoris and / or myocardial infarction within the 6 months prior to screening;
10. Subjects with concurrent or previously diagnosed with other malignancies, except for the patients under following conditions:

    * Well treated basal cells, papillary thyroid carcinoma, squamous cell carcinoma (adequate wound healing is required before enrollment into this study);
    * Carcinoma in situ of cervical cancer or breast cancer, after curative treatment, showed no signs of recurrence for at least 3 years before the study;
    * The primary malignancy has been completely removed and is in complete remission for 5 years.
11. Arrhythmic subjects without medical management control;
12. Subjects receiving oral anticoagulation within 1 week before JY231 injection infusion;
13. Having active neurological autoimmune or inflammatory conditions (such as Guillain-Barre syndrome, amyotrophic lateral sclerosis);
14. Female subjects in pregnant or lactating, or women with planned pregnancy within 2 years after JY231 infusion or male partner with planned pregnancy within 2 years after JY231 infusion;
15. Subjects with taboo study procedures or other medical conditions that may put them at unacceptable risk according to the investigator's judgment and / or clinical criteria.
16. Other conditions that the investigator believes that the subjects should not be enrolled in this clinical trial, such as poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events(AE) after infusion | Day 28、Month 2、Month 3、Month 6、Month 12、Month 18、Month 24
  The frequency, severity, and laboratory findings of all adverse events/serious adverse events are included.
Maximal Tolerated Dose(MTD) | Up to 28 days after infusion
  MTD will be determined based on Dose-Limiting Toxicity(DLTs) observed during the first 28 days of study treatment.

SECONDARY OUTCOMES:
Objective Response Rate | Day 28、Month 2、Month 3、Month 6、Month 12、Month 18、Month 24
  Objective Response Rate(ORR) is defined as the proportion of subjects achieving complete remission(CR) and partial response(PR)

CONTACTS AND LOCATIONS:
Overall Officials: Jia Wei, Doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, China, Wuhan, Hubei, China